CLINICAL TRIAL: NCT06239064
Title: Whole Genetic Approach in Early Genetic Identification of Obesity (WEGIO)
Brief Title: Early Genetic Identification of Obesity
Acronym: WEGIO
Status: Active, not recruiting | Type: Observational
Sponsor: Rolfs Consulting und Verwaltungs-GmbH (RCV) (Network)
Collaborators: Rhythm Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: WEGIO 01-2023
Record Dates: First submitted 2024-01-25; First posted 2024-02-02 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-02

CONDITIONS: Obesity, Childhood; Hyperphagia; Retinopathy; Syndactyly; Polydactyly; Cognitive Impairment; Bardet-Biedl Syndrome; POMC Deficiency
Keywords: Early onset obesity; Hyperphagia; Genetics; Bardet-Biedl Syndrome; LEPR; POMC; PCSK1
MeSH Terms: conditions — Pediatric Obesity; Hyperphagia; Retinal Diseases; Syndactyly; Polydactyly; Cognitive Dysfunction; Bardet-Biedl Syndrome; Proopiomelanocortin Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants suspected to genetic obesity: Participants suspected to genetic obesity
  Interventions: Diagnostic Test: Genetic testing via blood collection

INTERVENTIONS:
Diagnostic Test: Genetic testing via blood collection — blood collection

SUMMARY:
TITLE: Whole genetic approach in Early Genetic Identification of Obesity (WEGIO)

DESIGN: Multicenter epidemiological study

STUDY POPULATION: Participants at risk for a syndromic or a monogenic genetic obesity, incl. participants clinically diagnosed with Bardet-Biedl-Syndrome (BBS)

NUMBER OF PARTICIPANTS: 1000 for initial genetic sequencing and app. 40 for the follow-up documentation

COORDINATING INVESTIGATOR: Prof. Dr. Arndt Rolfs

DETAILED DESCRIPTION:
TITLE: Whole genetic approach in Early Genetic Identification of Obesity (WEGIO)

DESIGN: Multicenter epidemiological study

STUDY POPULATION: Participants at risk for a syndromic or a monogenic genetic obesity, incl. participants clinically diagnosed with Bardet-Biedl-Syndrome (BBS)

NUMBER OF PARTICIPANTS: 1000 for initial genetic sequencing and app. 40 for the follow-up documentation

COORDINATING INVESTIGATOR: Prof. Dr. Arndt Rolfs

PARTICIPATING COUNTRY: Germany

TREATMENT: Not applicable

PRIMARY OBJECTIVE: To investigate the prevalence of BBS in an at-risk population

SECONDARY OBJECTIVES:

* To explore genotype-phenotype correlation
* To assess genotypes distribution in Germany and compare to other countries
* To identify new genes/variants
* To investigate clinical characteristics in individuals diagnosed with BBS

DURATION OF RECRUITMENT: 32 months - total

24 months the recruitment of 1000 subjects

27 months follow up visits

32 months close out of sites

INCLUSION CRITERIA:

* Informed consent is obtained from the participant/parent/legal guardian
* The participant is 2 years of age or older

For a participant between 2 and 18 years of age:

* The participant has and had a body weight more than 97th percentile before the age of 6
* The participant has one or more of the following symptoms:

rod/cone dystrophy, renal abnormalities, ataxia, syndactyly, polydactyly, brachydactyly, hyperphagia, cognitive impairment, speech delay, hypogonadism

For a participant who is 18 years of age or older:

* The participant has BMI ≥ 30 kg/m2
* The participant had a body weight more than 97th percentile before the age of 6 years
* The participant has rod/cone dystrophy
* The participant is 2 or more years of age, is clinically diagnosed with Bardet-Biedl-Syndrome (BBS) or is a sibling of an individual diagnosed with BBS via the WEGIO study

ELIGIBILITY:
Inclusion criteria:

* Informed consent is obtained from the participant/parent/legal guardian
* The participant is 2 years of age or older

For a participant between 2 and 18 years of age:

* The participant has and had a body weight more than 97th percentile before the age of 6
* The participant has one or more of the following symptoms:

rod/cone dystrophy, renal abnormalities, ataxia, syndactyly, polydactyly, brachydactyly, hyperphagia, cognitive impairment, speech delay, hypogonadism

For a participant who is 18 years of age or older:

* The participant has BMI ≥ 30 kg/m2
* The participant had a body weight more than 97th percentile before the age of 6 years
* The participant has rod/cone dystrophy
* The participant is 2 or more years of age, is clinically diagnosed with Bardet-Biedl-Syndrome (BBS) or is a sibling of an individual diagnosed with BBS via the WEGIO study

Exclusion criteria:

- Not fulfilling the inclusion criteria

Min Age: 2 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Participants at risk for a syndromic or a monogenic genetic obesity, incl. participants clinically diagnosed with Bardet-Biedl-Syndrome (BBS)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
BBS prevalence | 2 years
  To investigate the prevalence of BBS in patients suspected to a genetic obesity

SECONDARY OUTCOMES:
Phenotypic and genetic characterization | 2 years
  To understand the genotype-phenotype correlation; to assess genotypes distribution in Germany and compare to other countries; to identify new genes/variants; to investigate clinical characteristics in individuals diagnosed with BBS

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Rolfs, PhD, MD, Study Chair — Rolfs Consulting und Verwaltungs-GmbH (RCV)
Locations (37):
- Germany (37):
  - Universitätsklinikum Aachen (RWTH), Aachen
  - KJF Klinik Josefinum, Augsburg
  - Universitätsklinikum Augsburg - Klinik für Kinder- und Jugendmedizin, Augsburg
  - Universitätsklinikum Freiburg, Bad Krozingen
  - Klinikum Bielefeld Mitte, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Praxis für Endokrinologie Dr. Daniel Pfaff, Bückeburg
  - Cellitinnen-Krankenkaus St. Franziskus, Cologne
  - Universitätsmedizin Essen, Essen
  - Klinikum Frankfurt (Oder), Frankfurt (Oder)
  - SRH Wald-Klinikum Gera, Gera
  - Universitätsmedizin Göttingen - Klinik für Kinder- und Jugendmedizin, Göttingen
  - WolfartKlinik, Gräfelfing
  - Universitätsmedizin Greifswald - Klinik und Poliklinik für Innere Medizin A, Greifswald
  - Katholisches Kinderkrankenhaus WILHELMSTIFT, Hamburg
  - Kinder- und Jugendkrankenhaus Auf der Bult, Hanover
  - Hormonzentrum Heidelberg, Heidelberg
  - Kinder- und Jugendarztpraxis Nebras Mohammad, Iserlohn
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel
  - Sozialpädiatrisches Zentrum Leipzig, Leipzig
  - Universitätsmedizin Mannheim - Augenklinik, Mannheim
  - Städtische Kliniken Mönchengladbach - Elisabeth-Krankenhaus Rheydt, Mönchengladbach
  - Kinder- und Jugendarztpraxis Sulaiman Al Sawaf, Nettetal
  - Dietrich-Bonhoeffer-Klinikum, Neubrandenburg
  - Hausarztpraxis Rahman & Detho, Obertshausen
  - Sana Klinikum Offenbach, Offenbach
  - Kinderärzte am Leo, Pforzheim
  - Klinikum Ernst von Bergmann, Potsdam
  - Elblandklinikum Riesa, Riesa
  - GPR Klinikum Rüsselsheim, Rüsselsheim am Main
  - Kinder- und Jugendpraxis Dogan, Stuttgart
  - SRH Zentralklinikum Suhl GmbH, Suhl
  - Praxis für Kinder- und Jugendmedizin Dr. med. Tabea Tippelt, Velbert
  - Dreifaltigkeits-Krankenhaus Wesseling, Wesseling
  - Praxis für Kinder- und Jugendmedizin Seyfullah Gökce, Wiesbaden
  - Universitätsklinikum Würzburg - Medizinische Klinik und Poliklinik I, Würzburg

IPD SHARING:
Plan to Share IPD: No